CLINICAL TRIAL: NCT03841396
Title: A Phase IV, Randomised, Double-blind Study Comparing the Local Tolerability of Two Subcutaneous Heparins, Fraxiparine and Clexane, in Healthy Volunteers.
Brief Title: A Study Comparing the Local Tolerability of Two Subcutaneous Heparins in Healthy Volunteers.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aspen Global Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CSA-15-ASP-002
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Injection Site Reaction
MeSH Terms: conditions — Injection Site Reaction | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study was planned to be a replicated 3x3 Latin square design (5 replicates), each enrolled and randomised participant should have received a single sequence of subcutaneous injections of Placebo, Fraxiparine and Clexane, in randomised order, on three separate occasions.
Who Masked: Participant, Investigator
Masking Description: This was a double blind study and it was conducted under double blind conditions. The study medications, as well as the placebo, were contained in pre-packaged syringes which are different in physical appearance. Therefore to ensure double blinding conditions, the study medications (Fraxiparine, Clexane and Placebo) were packaged in an identical boxes and labelled identically (apart from the treatment number). To further ensure that the participants remained blinded during the study, a blindfold was put over the eyes of each participant at each visit that required IP administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fraxiparine (Active Comparator): Nadroparine, Pre-filled syringe, 3800IU, single dose
  Interventions: Drug: Sodium chloride
- Clexane (Active Comparator): Enoxaparin, Pre-filled syringe, 40 mg, single dose
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium chloride — All participants received a single dose of sodium chloride as placebo
  Other Names: Saline 0.4mL saline

SUMMARY:
A Phase IV, Randomised, Double-blind, Single-centre clinical trial in healthy male and female participants aged 18 to 55, that was designed to assess and compare the pain intensity at an injection site as well as the duration of pain following a single dose subcutaneous administration of two low molecular weight heparins (LMWH) respectively.

DETAILED DESCRIPTION:
This was a Phase IV, Randomised, Double-blind, Single-centre clinical trial in healthy male and female participants aged 18 to 55, that was designed to assess and compare the pain intensity at an injection site as well as the duration of pain following a single dose subcutaneous administration of two LMWHs respectively. This study included an approximate seven-day screening period (screening visit to day 0), followed by three visits (Visit 2, 3 and 4) in one-week intervals, in which each participant should have received a single sequence of subcutaneous injections of Placebo, Fraxiparine and Clexane, in a randomised order, on the three separate occasions. This was then followed by a safety follow-up visit, one week after the administration of the last dose of the study product.

Fifteen (N = 15) healthy, consenting participants, fulfilling the inclusion criteria, were randomised to take part in this study. All participants received a single sequence of subcutaneous injections, on separate occasions at one week intervals, over the duration of the treatment phase of the study. Fifteen (N=15) participants received Fraxiparine, fifteen (N=15) participants received Clexane and fifteen (N=15) participants received Placebo. Two participants were screened however did not meet the eligibility criteria and therefore were not included into the study. Informed consent was obtained at Screening Visit 1 (day -7 to 0) before any trial-related procedures were be performed. Visual analogue and 11-point numeric rating scales were utilised to measure pain intensity after a single injection of investigational product. These scales were also used to assess burning and pruritus. All scales were be completed at set time intervals over a 30 minute period, i.e. 1, 3, 5, 10, 15 and 30 minutes after the injections were completed. Hematoma, erythema and oedema were measured minutes and 1, 2 and 3 days after the injection, using transparent millimetric measuring paper. Safety bloods were drawn at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female participant.
2. Aged 18 years to 55 years.
3. Medically healthy participants.
4. Weight Females: ≥ 45 kg; Males ≥ 57 kg.
5. Body Mass Index (BMI) of 18,5 to 29,9 kg/m2.
6. Female participants of child-bearing potential must have a negative urine pregnancy test at screening and be willing to use effective contraceptives throughout the trial duration.
7. Participants must be able to understand and follow the instructions of the Investigator, understand and give informed consent, and be willing, committed, and able to return for all site visits and complete all study-related procedures.

Exclusion Criteria:

1. A known hypersensitivity to Clexane or Fraxiparine or any components thereof - especially allergies to latex, pork products, sulfites and benzyl alcohols.
2. Female participants who are pregnant or lactating.
3. Any coagulopathy - Anaemia, thrombocytopenia, hemophilia, haemorrhagic diathesis (Bleeding, Bruising, Clotting disorders).
4. Active gastric or duodenal ulcer or history of previous gastric duodenal bleeding or gastrointestinal bleeding.
5. Participants on the following medications: Anti-coagulants, Non-Steroidal Anti-inflammatory Drugs (NSAID)s, glycoprotein IIb/IIIa anticoagulants, thrombolytic agents, platelet-inhibitors, acetylsalicylic acid, sulfinpyrazone, quinine - containing remedies and/drinks, treprostinil, apixaban, drotecogin alfa, danshen, dong quai, evening primrose oil, gingko, policosanol and willow bark as well as hyperkalemia aggravators in the last 7 days.
6. A Cerebrovascular incident (hemorrhagic or ischemic).
7. Deep Vein Thrombosis and/ Pulmonary embolism.
8. Acute infective endocarditis or history of acute endocarditis.
9. Participants with Hypertension.
10. Diabetics.
11. Any injuries or surgery of the ears, eyes, brain or spinal cord within the last 18 months.
12. Renal insufficiency (Creatinine and Urea not within normal ranges).
13. Hepatic Insufficiency ( aspartate aminotransferase (AST) and alanine transaminase (ALT) within normal ranges).
14. Participants with Heamorrhagic Retinopathy.
15. Participants with prosthetic heart valve/s.
16. Participants currently receiving any other treatments administered via subcutaneous or intramuscular routes.
17. Participants with a history or current endocrine, pulmonary, cardiovascular, gastrointestinal, neurological, immunological, renal, hepatic, dermatologic, haematologic, psychiatric disease other than specified that might have/cause unwanted effects/outcomes in this clinical trial.
18. Alcohol and/ or drug abuse in the past year.
19. In the opinion of the investigator, the participant is not reliable to participate in the trial.
20. Participants that have taken part in a clinical trial involving Clexane and/ Fraxiparine.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Comparison of Visual Analog Scale (VAS) scores of pain intensity at injection site following a single subcutaneous injection of placebo, Fraxiparine or Clexane | Over a period of 30 minutes
  Visual Analogue Scales for pain intensity was performed at different time points namely 1, 3, 5, 10, 15 and 30 minutes after administration of the investigational product (IP) at Visit 2, 3 and 4. Pain intensity: 0 mm - No pain; 100 mm - Worst pain
Comparison of Numeric Rating Scale (NRS) scores of pain intensity at injection site following a single subcutaneous injection of placebo, Fraxiparine or Clexane. | Over a period of 30 minutes
  11-point NRS for pain intensity was performed at different time points namely 1, 3, 5, 10, 15 and 30 minutes after administration of the investigational product (IP) at Visit 2, 3 and 4. Pain intensity: 0 - No pain; 10 - Worst pain

SECONDARY OUTCOMES:
Quantification of local injection site reaction | 10 and 30 minutes and 1, 2 and 3 days after the injection.
  Hematoma, erythema and oedema were measured 10 and 30 minutes and 1, 2 and 3 days after the injection, using transparent millimetric measuring paper.
Pain duration | 1, 3, 5, 10, 15 and 30 minutes after administration of IP.
  Duration of pain at injection site.

IPD SHARING:
Plan to Share IPD: No